CLINICAL TRIAL: NCT00516464
Title: Evaluation of Ranibizumab on the Ease of Procedure and Complication Rate in Proliferative Diabetic Retinopathy (PDR) Requiring Vitrectomy
Brief Title: Evaluation of Ranibizumab in Proliferative Diabetic Retinopathy (PDR) Requiring Vitrectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Retina Associates, Kansas City (Other)
Collaborators: Genentech, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: FVF4295
Record Dates: First submitted 2007-08-14; First posted 2007-08-15 (Estimated); Last update posted 2007-08-15 (Estimated); Status verified 2007-08

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: Proliferative Diabetic Retinopathy; Vitrectomy; Ranibizumab
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Lucentis (ranibizumab)

SUMMARY:
Evaluation of ranibizumab on the ease and procedure and complication in proliferative diabetic retinopathy (PDR) requiring vitrectomy.

DETAILED DESCRIPTION:
This is an open-label, Phase I/II study of multiple doses of intravitreally administered ranibizumab in patients with severe NPDR and PDR prior to, during, and after vitrectomy therapy.

40 subjects will be enrolled and randomized 3:1 to ranibizumab or vitrectomy alone. 30 consented, enrolled subjects will receive 3 intravitreal injections of 0.5 mg ranibizumab administered 1-3 weeks pre-procedure, intraoperatively, and 1 month post-vitrectomy.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 20 years
* Best corrected visual acuity of 20/40 to 20/800 in the study eye
* Very servere nonproliferative diabetic retinopathy (ETDRS level 53E) OR moderate proliferative diabetic retinopathy (ETDRS level 65)
* Visual reduction attributable to diabetic vitreous hemorrhage or diabetic macular edema
* Candidate for vitrectomy procedure

Exclusion Criteria:

* Pregnancy (positive Pregnancy test) or lactation
* Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated.
* Participation in another simultaneous medical investigation or trial.
* Visual impairment attributable to causes other than diabetic macular edema or diabetic vitreous hemorrhage.
* Use of intraocular or periocular corticosteroids within 6 months.
* History of panretinal photocoagulation
* History of macular laser photocoagulation
* History of pars plana vitrectomy
* Prior or concomitant treatment with ranibizumab, bevacizumab, or pegaptanib sodium, either as part of an investigational study or as an off-label medication.
* Current treatment of a systemic infection

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-08; Study Completion 2008-08 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of ranibizumab on vitrectomy complications such as recurrent vitreous hemorrhage, postoperative retinal detachment rates, and development of intraoperative retinal breaks. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gregory M Fox, MD, Principal Investigator — Retina Associates, PA
Locations (1):
- Retina Associates, PA, Shawnee Mission, Kansas, United States

REFERENCES:
- [Derived] Dervenis P, Dervenis N, Smith JM, Steel DH. Anti-vascular endothelial growth factors in combination with vitrectomy for complications of proliferative diabetic retinopathy. Cochrane Database Syst Rev. 2023 May 31;5(5):CD008214. doi: 10.1002/14651858.CD008214.pub4. PMID 37260074